CLINICAL TRIAL: NCT00768339
Title: AEG35156-204: A Phase 1-2, Multicenter, Open-Label Study of the X-Linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia and Indolent B-Cell Lymphomas
Brief Title: A Phase 1-2, Multicenter, Open-Label Study of AEG35156 in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia and Indolent B-Cell Lymphomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Aegera Therapeutics (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-204
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell
Keywords: antisense; AEG35156; lymphocytic; lymphoma; leukemia; B-cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single agent AEG35156 as 2hr IV infusion, weekly dosing in Patients with relapsed or refractory chronic lymphocytic leukemia and indolent B-cell lymphomas
  Interventions: Drug: AEG35156 antisense IV infusion

INTERVENTIONS:
Drug: AEG35156 antisense IV infusion — AEG35156 will be given as a 2-hour intravenous infusion (escalating dose 50, 100, 150, 200, 250 and 300 mg) once weekly on Day 1, Day 8 and Day 15. One cycle of therapy will consist of 21 days. Patients will be treated until disease progression.
  * Patients must be pretreated for at least three days with allopurinol prior to the first dose of AEG35156 and throughout protocol therapy.
  * Patients must be hydrated with 1 L of normal saline prior AEG35156 infusion
  Other Names: XIAP antisense

SUMMARY:
AEG35156 has shown early evidence of activity in patients with advanced indolent B-cell lymphomas in Phase 1 trials and merits further evaluation in this disease. This trial is designed to determine the recommended dose of AEG35156 in patients with relapsed or refractory chronic lymphocytic leukemia (CLL) and indolent B-cell lymphomas.

DETAILED DESCRIPTION:
Apoptotic induction in cancer cells is a sought after therapeutic goal. Most successful anticancer agents activate apoptosis pathways in the cancers they treat. Apoptotic pathways in cells appear to converge on a single family of enzymes, the caspases, which are proteases that dismantle the cell in an orderly, non-inflammatory fashion, resulting in cell death. The X-linked Inhibitor of Apoptosis (XIAP) is the only known cellular inhibitor of caspases, its over expression thereby blocking the principal means of apoptosis. A wide range of evidence indicates that cellular overexpression of members of the IAP family is a fundamental means by which many cancer cells evade death, even in the presence of strong extrinsic (death receptor-mediated) and intrinsic (mitochondria-mediated) apoptotic cues. The inhibition of cellular XIAP activity, specifically in cancer cells under stress and primed for apoptosis by chemotherapeutic agents, is viewed as a powerful means of tipping the balance towards cell death. In particular, XIAP has been shown to be overexpressed in lymphoma. AEG35156 is a second generation antisense which targets XIAP mRNA to lower XIAP levels and the apoptotic threshold of cancer cells, enhancing their sensitivity to intrinsic death and chemotherapy. AEG35156 has shown early evidence of activity in patients with advanced indolent B-cell lymphomas in Phase 1 trials and merits further evaluation in this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an histologically confirmed diagnosis of CLL as per NCI-WG criteria or
* Patients with an histologically confirmed diagnosis of one of the following indolent B-cell lymphomas: (Follicular lymphoma (FL); Small lymphocytic lymphoma (SLL); Marginal zone lymphoma; Lymphoplasmacytic lymphoma)
* Relapsed or refractory patients who have failed at least 2 prior lines of therapy, one of which may have been high dose therapy and autologous stem cell transplantation. Steroids alone when used for autoimmune phenomena do not qualify as prior therapy
* ECOG performance less or equal than 2
* Life expectancy of at least 3 months
* Age greater or equal than 18 years
* Signed, written IRB-approved informed consent
* A negative serum pregnancy test (if applicable)
* Acceptable liver function:(Bilirubin within normal limit; AST (SGOT) and ALT (SGPT) less or equal than 2.5 x ULN or less or equal than 5 x ULN if there are liver lymphomatous involvement)
* Acceptable renal function: (Serum creatinine within normal limits, OR calculated creatinine clearance greater or equal than 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal)
* Acceptable hematologic status: (Granulocyte greater or equal than 1000 cells/uL; Platelet count greater or equal than 50,000 /uL)
* Acceptable coagulation status:(PT within normal limits; PTT within normal limits)
* For women of child-producing potential, the use of effective contraceptive methods during the study
* Prior radiotherapy for local disease is allowed provided disease progression has been documented, and treatment completed at least 4 weeks prior to registration

Exclusion Criteria:

* Uncontrolled autoimmune hemolysis and/or thrombocytopenia
* Richter's transformation
* Histologic transformation
* Patients with peripheral neuropathy
* Active progressive leptomeningeal disease including the presence of any related symptoms or need for corticosteroids. A CT or MRI scan of the head is necessary in patients with a history of leptomeningeal disease to document the stability of prior lesions
* Pregnant or nursing women. NOTE: Women of child-bearing potential must agree to use adequate contraception (sterile or surgically sterile; hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Men who are unwilling to use acceptable forms of birth control when engaging in sexual contact with women of child bearing potential
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent. Subjects who have used a previous antisense oligonucleotide in the last 90 days will be excluded
* Unwillingness or inability to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response according to CLL NCI-WG criteria | Every numbered cycles

CONTACTS AND LOCATIONS:
Overall Officials: John Sweetenham, MD, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (4):
  - Providence Saint-Joseph Medical Center, Burbank, California
  - New York Medical College, Valhalla, New York
  - The Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - Scott and White Memorial Hospital, Temple, Texas
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital - Sir Mortimer B. Davis, Montreal, Quebec